CLINICAL TRIAL: NCT04825171
Title: Perceived Changes in Anxiety Symptom Burden During Treatment With Bryophyllum Pinnatum and Tolerability: a Prospective, Single-Group Pre-post Observational Study as Investigator-Initiated Trial (IIT)
Brief Title: Perceived Changes in Anxiety Symptom Burden During Treatment With Bryophyllum Pinnatum and Tolerability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Markus Schlemmer (Other)
Responsible Party: Sponsor-Investigator, Markus Schlemmer, Dr. med., Klinik Arlesheim
Organization: Klinik Arlesheim (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bryo-KLA-02
Record Dates: First submitted 2021-03-15; First posted 2021-04-01 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Anxiety Symptoms
Keywords: Anxiety; Depression; Stress; Sleep Quality; Internal Coherence
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders | interventions — Mastication; lipoarabinomannan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bryophyllum pinnatum 50% chewing tablets (Experimental): Bryophyllum is administered for 3 weeks. Bryophyllum is given in form of chewing tablets, 350mg per tablet, 0-2-2-2/d: 2 tablets at midday, 2 tablets in the evening, 2 tablets before bedtime.
  Interventions: Drug: Bryophyllum 50 % Chewing Tablets

INTERVENTIONS:
Drug: Bryophyllum 50 % Chewing Tablets — Each 350 mg tablet corresponds to 170 mg of leave press juice from Bryophyllum pinnatum, dried down to 17 mg by mixing with lactose; 100 mg dried BP matter in 1 g.
  Other Names: Bryophyllum pinnatum/Kalanchoe, Bryophyllum pinnatum (Lam.) Oken.

SUMMARY:
Bryophyllum pinnatum (BP) is a succulent perennial plant from the family Crassulacea (for reviews see Fürer 2016 and Hamburger 2017). Leaf extracts from BP have been used in traditional medicine to treat wounds and ulcers, skin diseases, infections, inflammations, pain, diabetes, hypertension, and cancer. In Europe, BP started to be used at the beginning of the 20th century in Anthroposophic medicine, a form of holistic medicine with an integrative approach. Almost a hundred years later, BP preparations are still often prescribed in Anthroposophic medicine, where it is used in the treatment of a broad spectrum of diagnoses, most often of mental and behavioural disorders (ICD-10 F00-F99), including anxiety, depressive, and sleep disorders (Simões-Wüst 2012).

In Switzerland, during the last decade, BP (50 % tablets) started to be used in conventional settings mainly in the treatment of preterm labour (Simões-Wüst 2018, Plangger 2006), overactive bladder (Betschart 2013), sleep disorders (Simões-Wüst 2015), and restless legs syndrome (Von Manitius 2019).

Whereas the good effectiveness of BP preparations in the treatment of preterm contractions and overactive bladder is well supported by data obtained using a variety of in vitro models (see e.g. Santos 2018, Bachmann 2017, Simões-Wüst 2010), less is known about possible mechanisms of action that would support their use in the treatment of mental and behavioural disorders.

Nevertheless, the observed improvements of sleep disorders are corroborated by animal experiments showing that different fractions of the leaf extract of BP can prolong the pentobarbitone-induced sleeping time (Yemitan 2005 and Pal 1999), indicating a CNS depressant action. Some of the bufadienolides present in Bryophyllum species are thought to be responsible for the sedative effects (Wagner 1986).

The aim of the present study is to find out if patients suffering from anxiety symptoms perceive improvements of these symptoms during treatment with Bryophyllum 50% tablets. Since anxiety symptoms are often related to depression, reduced sleep quality, stress, reduced health-related quality of life and the feeling of not being able to control owns life (internal coherence), these aspects will be assessed as well.

DETAILED DESCRIPTION:
The present IIT (Investigator-Initiated Trial) study is a prospective, single-group, pre-post study (phase IV).

A past study showed that among Anthroposophical physicians the most frequent diagnosis group where BP preparations are prescribed are mental and behavioural disorders such as anxiety and sleep disorders. In the present study, we, therefore, want to investigate the effectiveness of Bryophyllum tablets in patients with anxiety symptoms.

Study participants will be recruited among the patients on the waiting list of the Department of Psychiatry and Psychosomatics at the Clinic Arlesheim.

* Participant recruitment will continue until 60 patients have concluded the study.
* Recruitment period will probably last 15 months.
* Duration of the drug administration is 3 weeks.

Participants will fill in a questionnaire three times. At baseline, after two and after three weeks of Bryophyllum intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred by their treating physician to the Department of Psychiatry and Psychosomatic of the Clinic Arlesheim waiting for the in-stay
* Expected waiting time until in-stay is at least two weeks
* Patients having anxiety symptoms as measured by the GAD-2 questionnaire (cut-off of 3 points)
* Patients'state of health allows them to complete the questionnaire on their own
* Signed informed consent
* No treatment with BP during the last two months
* No planned doses increase of (conventional) anxiolytics or antidepressants for the duration of the period until in-stay
* Age over 18 years
* Good German knowledge (at least level B2 from Common European Framework of Reference for Languages)

Exclusion Criteria:

* Wheat allergies
* Acute life-threatening conditions
* Withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change of anxiety symptoms | 2 weeks
  Assessed with the Beck Anxiety Inventory (BAI, Beckler 2010) score between before treatment and after 2 weeks of treatment. BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults. The questions ask about common symptoms of anxiety that the subject has had during the past week (including the day you take it) (such as numbness and tingling, sweating not due to heat, and fear of the worst happening). Each answer to a BAI-question is scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cut-offs are: 0-7, minimal anxiety; 8-15, mild anxiety; 16-25, moderate anxiety; 26-63, severe anxiety.

SECONDARY OUTCOMES:
Change of anxiety symptoms | 3 weeks
  Assessed with the Beck Anxiety Inventory (BAI) score between before treatment and after 3 weeks of treatment.
Change of anxiety symptoms | 2 and 3 weeks
  Assessed with the Generalized Anxiety Disorder (GAD-7, Williams 2014) questionnaire. GAD-7 is used to measure symptoms and severity of anxiety; scores range from 0 to 21, with higher scores indicating more severe symptoms. Total scores classify symptoms as normal (0-4), mild (5-9), moderate (10-14), and severe (15-21). A total score≥8 is indicative of clinically significant anxiety symptoms.
Change of depression symptoms | 2 and 3 weeks
  Assessed with the nine-question depression scale (PHQ-9, Spitzer 1999). PHQ-9 is used to assess the presence and severity of depressive symptoms; scores range from 0 to 27, with higher scores indicating more severe symptoms. Total scores classify depression symptoms as normal (0-4), mild (5-9), moderate (10-14), moderate-severe (15-19) and severe (20-27). A total score ≥10 is indicative of clinically significant symptoms of depression and of a DSM-IV diagnosis of depression.
Change of stress symptoms | 2 and 3 weeks
  Assessed with the Perceived Stress Scale (PSS, Klein 2016). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Change in sleep quality | 2 and 3 weeks
  Assessed with the Pittsburgh Sleep Quality Index (PSQI, Buysse 1989). The PSQI contains 19 self-rated questions and are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score o "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
Change in health-related quality of life questionnaire | 2 and 3 weeks
  Assessed with the Health-related Quality of Life questionnaire (SF-12, Morfeld 2011). The 12 items allow the calculation of two health summary measures, namely physical health summary and mental health summary scales. The scores range from 0 to 60 with higher scores indicating higher degree of difficulty in life.
Change in the Sense of Coherence | 2 and 3 weeks
  Assessed with the Internal Coherence Scale (ICS, Kröz 2009). The scores range from 1-50 with higher scores indicating higher degree of internal coherence.
Brophyllum Prescription report | 3 weeks
  It is examined whether and which participants asked for a Bryophyllum 50 % prescription after the study.

OTHER OUTCOMES:
Incidence of any Adverse Events (Safety) | 2 and 3 weeks
  All perceived events and side effects are recorded by the participant in the questionnaires and any SAE is reported to the study team by telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schlemmer, Dr. med., Principal Investigator — Klinik Arlesheim, Pfeffingerweg1, 4144 Arlesheim, Switzerland
Locations (1):
- Klinik Arlesheim, Arlesheim, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication can be shared with other researchers.
Supporting Information: ICF
Time Frame: IPD and additional supporting information will become available 6 months after publication for 6 months.
Access Criteria: Additional information can be gained on request. We then decide whether we want to share additional data or not.

REFERENCES:
- [Background] Furer K, Simoes-Wust AP, von Mandach U, Hamburger M, Potterat O. Bryophyllum pinnatum and Related Species Used in Anthroposophic Medicine: Constituents, Pharmacological Activities, and Clinical Efficacy. Planta Med. 2016 Jul;82(11-12):930-41. doi: 10.1055/s-0042-106727. Epub 2016 May 24. PMID 27220081
- [Background] M. Hamburger, O. Potterat, K. Fürer, A. P. Simões-Wüst, and U. Von Mandach, "Bryophyllum pinnatum - Reverse engineering of an anthroposophic herbal medicine," in Natural Product Communications, 2017, vol. 12, no. 8, pp. 1359-1364.
- [Background] Simoes-Wust AP, Lapaire O, Hosli I, Wachter R, Furer K, Schnelle M, Mennet-von Eiff M, Seifert B, von Mandach U. Two Randomised Clinical Trials on the Use of Bryophyllum pinnatum in Preterm Labour: Results after Early Discontinuation. Complement Med Res. 2018;25(4):269-273. doi: 10.1159/000487431. Epub 2018 Jun 22. No abstract available. PMID 29945146
- [Background] Betschart C, von Mandach U, Seifert B, Scheiner D, Perucchini D, Fink D, Geissbuhler V. Randomized, double-blind placebo-controlled trial with Bryophyllum pinnatum versus placebo for the treatment of overactive bladder in postmenopausal women. Phytomedicine. 2013 Feb 15;20(3-4):351-8. doi: 10.1016/j.phymed.2012.10.007. Epub 2012 Dec 4. PMID 23218404
- [Background] Schenkel L, Simoes-Wust AP, Hosli I, von Mandach U. Drugs in Pregnancy and Lactation - Medications Used in Swiss Obstetrics. Z Geburtshilfe Neonatol. 2018 Feb 8. doi: 10.1055/s-0043-124975. Online ahead of print. PMID 29421836
- [Background] Furer K, Simoes-Wust AP, Winkler A, Amsler N, Schnelle M, von Mandach U. [The Application of Bryophyllum pinnatum Preparations in Obstetrics and Gynaecology - a Multicenter, Prospective Observational Study]. Forsch Komplementmed. 2015;22(4):231-6. doi: 10.1159/000437154. Epub 2015 Aug 3. German. PMID 26228703
- [Background] Santos S, Haslinger C, Klaic K, Faleschini MT, Mennet M, Potterat O, von Mandach U, Hamburger M, Simoes-Wust AP. A Bufadienolide-Enriched Fraction of Bryophyllum pinnatum Inhibits Human Myometrial Contractility In Vitro. Planta Med. 2019 Mar;85(5):385-393. doi: 10.1055/a-0810-7704. Epub 2018 Dec 18. PMID 30562827
- [Background] Pal S, Sen T, Chaudhuri AK. Neuropsychopharmacological profile of the methanolic fraction of Bryophyllum pinnatum leaf extract. J Pharm Pharmacol. 1999 Mar;51(3):313-8. doi: 10.1211/0022357991772312. PMID 10344633
- [Background] Yemitan OK, Salahdeen HM. Neurosedative and muscle relaxant activities of aqueous extract of Bryophyllum pinnatum. Fitoterapia. 2005 Mar;76(2):187-93. doi: 10.1016/j.fitote.2004.11.009. PMID 15752629
- [Background] H. Wagner, H. Lotter, and M. Fischer, "Die toxischen und sedierend wirkenden Bufadienolide von Kalanchoedaigremontiana HAMETet PERR," Helv. Chim. Acta, vol. 69, no. 2, pp. 359-367, 1986.
- [Background] Furer K, Raith M, Brenneisen R, Mennet M, Simoes-Wust AP, von Mandach U, Hamburger M, Potterat O. Two new flavonol glycosides and a metabolite profile of Bryophyllum pinnatum, a phytotherapeutic used in obstetrics and gynaecology. Planta Med. 2013 Nov;79(16):1565-71. doi: 10.1055/s-0033-1350808. Epub 2013 Sep 26. PMID 24072500
- [Background] Plangger N, Rist L, Zimmermann R, von Mandach U. Intravenous tocolysis with Bryophyllum pinnatum is better tolerated than beta-agonist application. Eur J Obstet Gynecol Reprod Biol. 2006 Feb 1;124(2):168-72. doi: 10.1016/j.ejogrb.2005.05.013. Epub 2005 Jul 26. PMID 16051414
- [Background] Simoes-Wust AP, Jeschke E, Mennet M, Schnelle M, Matthes H, von Mandach U. Prescribing pattern of Bryophyllum preparations among a network of anthroposophic physicians. Forsch Komplementmed. 2012;19(6):293-301. doi: 10.1159/000345841. Epub 2012 Dec 17. PMID 23343584
- [Background] Lambrigger-Steiner C, Simoes-Wust AP, Kuck A, Furer K, Hamburger M, von Mandach U. Sleep quality in pregnancy during treatment with Bryophyllum pinnatum: an observational study. Phytomedicine. 2014 Apr 15;21(5):753-7. doi: 10.1016/j.phymed.2013.11.003. Epub 2013 Dec 25. PMID 24373544
- [Background] Simoes-Wust AP, Hassani TA, Muller-Hubenthal B, Pittl S, Kuck A, Meden H, Eberhard J, Decker M, Furer K, von Mandach U; Bryophyllum Collaborative Group. Sleep Quality Improves During Treatment With Bryophyllum pinnatum: An Observational Study on Cancer Patients. Integr Cancer Ther. 2015 Sep;14(5):452-9. doi: 10.1177/1534735415580680. Epub 2015 Apr 14. PMID 25873294
- [Background] von Manitius S, Flugel D, Gievers Steinlein B, Schnelle M, von Mandach U, Simoes-Wust AP. Bryophyllum pinnatum in the treatment of restless legs syndrome: A case series documented with polysomnography. Clin Case Rep. 2019 Apr 14;7(5):1012-1020. doi: 10.1002/ccr3.2144. eCollection 2019 May. PMID 31110737
- [Background] K. Beckler, "State-Trait Anxiety Inventory for Adults - Manual, Instrument and Scoring Guide," 1983 Consult. Psychol. Press. Inc. Mind Gard. Inc., pp. 0-78, 2010.
- [Background] N. Williams, "The GAD-7 questionnaire," Occup. Med. (Chic. Ill)., vol. 64, no. 3, p. 224, 2014.
- [Background] R. L. Spitzer, K. Kroenke, and J. B. W. Williams, "Validation and utility of a self-report version of PRIME-MD," Prim. Care Companion J. Clin. Psychiatry, vol. 2, no. 1, p. 31, 1999.
- [Background] Klein EM, Brahler E, Dreier M, Reinecke L, Muller KW, Schmutzer G, Wolfling K, Beutel ME. The German version of the Perceived Stress Scale - psychometric characteristics in a representative German community sample. BMC Psychiatry. 2016 May 23;16:159. doi: 10.1186/s12888-016-0875-9. PMID 27216151
- [Background] M. Morfeld, I. Kirchberger, and M. Bullinger, SF-36 Fragebogen zum Gesundheitszustand: Deutsche Version des Short Form-36 Health Survey. Hogrefe, 2011.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771